CLINICAL TRIAL: NCT07168434
Title: A Double-blind, Randomized, Placebo-controlled, Multicenter Trial Evaluating the Efficacy and Safety of Saccharomyces Boulardii CNCM I-745 in Adult Patients With Non-constipated Irritable Bowel Syndrome
Brief Title: Saccharomyces Boulardii CNCM I-745 in Irritable Bowel Syndrome
Acronym: BoWell Sb252
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Biocodex (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BoWell Sb252; 2024-520276-10-00 (EU CTIS Number)
Record Dates: First submitted 2025-08-22; First posted 2025-09-11 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: IBS (Irritable Bowel Syndrome); IBS-D (Diarrhea-predominant); IBS, Mixed Symptoms
Keywords: IBS; Irritable Bowel Syndrome; Saccharomyces boulardii; Non-constipated IBS
MeSH Terms: conditions — Irritable Bowel Syndrome; Ichthyosis Bullosa of Siemens

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment (Experimental): Saccharomyces boulardii CNCM I-745, 250 mg, 2 capsules/day
  Interventions: Drug: Saccharomyces Boulardii 250 MG
- Placebo (Placebo Comparator): Placebo, 250mg, 2 capsules/day
  Interventions: Drug: Placebo 250 mg

INTERVENTIONS:
Drug: Saccharomyces Boulardii 250 MG — Saccharomyces boulardii CNCM I-745, 250 mg, 2 capsules/day
  Arms: Treatment
Drug: Placebo 250 mg — Placebo, 250mg, 2 capsules/day
  Arms: Placebo

SUMMARY:
This is a double-blind, randomized (group assignment by chance), placebo-controlled, multicenter trial which will be conducted over a 13.5-months period The main objective of the research is to demonstrate the efficacy of Saccharomyces boulardii CNCM I-745 on global IBS symptoms, measured by the Irritable Bowel Syndrome Symptom Severity Scale (IBS-SSS), in comparison to placebo after 8 weeks.

Secondary efficacy objectives are to evaluate the impact of Saccharomyces boulardii CNCM I-745 on quality of life of IBS patients and on global and individual IBS symptoms, using the IBS-SSS, in comparison to placebo at regular intervals over a 3-month treatment period. This research also aims to evaluate the proportion of patients who improved ≥ 50 points on IBS-SSS and the proportion of responders according to the European Medicines Agency (EMA) definition (based on the patient's global assessment of efficacy and on abdominal pain score), after 8 weeks of treatment. Secondary safety objective is to evaluate the safety profile and tolerability of Saccharomyces boulardii CNCM I-745 capsules 500 mg/day in IBS patients in comparison to placebo

ELIGIBILITY:
Inclusion Criteria:

1. Male or female aged ≥ 18 and ≤ 65 years.
2. Diagnosis of IBS of any subtype, except constipation predominant (IBS-C), according to Rome IV criteria.
3. IBS-SSS total score ≥ 175 at inclusion.
4. Able and willing to maintain their nutrition habits throughout the study participation.
5. Able to understand and willing to comply with study requirements and to provide written informed consent.
6. For women of childbearing potential: willing to use one or more acceptable birth control method throughout the study participation.

Exclusion Criteria:

1. Diagnosis of IBS-C according to Rome IV criteria.
2. Patient with more than 5 bowel movements per day on average during the screening period, according to the patient's diary (BSFS).
3. Severe illness(es) or medical condition(s), including gastrointestinal pathologies (other than IBS): gastrointestinal ulcers, coeliac disease, inflammatory bowel disease, bowel cancer, acute or chronic diarrhea secondary to confirmed infectious gastroenteritis, or enteral or parenteral nutrition.
4. History of abdominal surgery (except for appendectomy, cholecystectomy, surgery for hemorrhoids or cesarian section, more than 6 months prior to inclusion).
5. Familial colorectal cancer syndrome (Lynch, Familial Adenomatous Polyposis).
6. Fecal transplant within 6 months prior to screening.
7. Use of products marketed as prebiotics, probiotics or synbiotics within 2 weeks prior to screening. These products, with the exception of the investigational product, will not be allowed during the trial. Regular cheese or yogurt containing lactic acid bacteria are not an exclusion criterion.
8. Systemic antibiotic or antimycotic treatment within 2 weeks prior to randomization. These treatments are not allowed during the study.
9. Laxatives, antibloating agents, antidiarrheal medication, antispasmodics, within 2 weeks prior to screening. These treatments are not allowed during the study, except loperamide which can be used as rescue medication.
10. Daily or regular non-steroidal anti-inflammatory drugs (NSAIDS) at doses above cardiovascular prophylaxis (low dose aspirin) are not allowed within 2 weeks prior to screening and throughout the study participation.
11. Use of opioids or narcotic analgesics, including tramadol and codeine, within 6 weeks prior to screening. These treatments are not allowed during the study.
12. Treatment with two or more antidepressant/anxiolytic/antipsychotic within 3 months prior to study entry or during the trial. Treatment with a single antidepressant or anxiolytic or antipsychotic agent before and during the trial is allowed provided that the dose is stable within 3 months prior to study entry and during the trial participation.
13. Treatment with anticholinergics for overactive bladder such as solifenacin, darifenacin, oxybutynin, tolterodine, fesoterodin, propiverin, trospium chloride, or mirabegron, within 1 week prior to screening. These treatments are not allowed during the study.
14. Allergy to yeast, especially Saccharomyces boulardii, or known hypersensitivity to one of the components.
15. Patients having a central venous catheter, critically ill patients, and immunocompromised patients.
16. Patients with rare hereditary problems of galactose or fructose intolerance, total lactase deficiency, glucose-galactose malabsorption or sucrase-isomaltase insufficiency.
17. Excessive alcohol consumption (>7 units/week) and/or drug abuse.
18. Other medical conditions or comorbidities, treatment, which in the opinion of the investigator, would interfere with study compliance or data interpretation.
19. Presenting any significant biological or clinical anomalies that are not compatible with participation in the study according to the investigator.
20. Participant at risk of pregnancy, pregnant or breastfeeding female.
21. Participant under guardianship or curatorship.
22. Participant under the protection of the Court or deprived of liberty.
23. Participant participating in another interventional clinical trial which could interfere with the trial's results or impact the other trial's results; or within 5 half-lives of the study investigational treatment, whichever is longer.
24. Participant whose current state of health does not allow him/her to give consent.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 406 (Estimated)
Dates: Start 2025-10-22 (Actual); Primary Completion 2026-10-11 (Estimated); Study Completion 2026-10-11 (Estimated)

PRIMARY OUTCOMES:
To demonstrate the efficacy of Saccharomyces boulardii CNCM I-745 on global Irritable Bowel Syndrome (IBS) symptoms, measured by the Irritable Bowel Syndrome Symptom Severity Scale (IBS-SSS), in comparison to placebo after 8 weeks. | From baseline to day 56
  Irritable Bowel Syndrome Symptom Severity Scale (IBS-SSS) is a scale evaluating the severity of the disease from 0 (minimum score : not severe) to 500 (maximum score : severe).

SECONDARY OUTCOMES:
To evaluate the impact of Saccharomyces boulardii CNCM I-745 on quality of life of Irritable Bowel Syndrome (IBS) patients in comparison to placebo. | From baseline to day 56 and from baseline to day 84
  Absolute change measured in the Irritable Bowel Syndrome-Quality of Life (IBS-QOL). Minimum score is 0 : poor quality of life. Maximum score : 100 : better quality of life.
To demonstrate the efficacy of Saccharomyces boulardii CNCM I-745 on global and individual Irritable Bowel Syndrome (IBS) symptoms, measured by the Irritable Bowel Syndrome Symptom Severity Scale (IBS-SSS), at each time point, in comparison to placebo. | From baseline to day 28, day 56 and day 84
  Irritable Bowel Syndrome Symptom Severity Scale (IBS-SSS) is a scale evaluating the severity of the disease from 0 (minimum score : not severe) to 500 (maximum score : severe).
To evaluate the proportion of patients who improved ≥ 50 points on Irritable Bowel Syndrome Symptom Severity Scale (IBS-SSS). | At day 28, day 56 and day 84 compared with baseline
  Irritable Bowel Syndrome Symptom Severity Scale (IBS-SSS) is a scale evaluating the severity of the disease from 0 (minimum score : not severe) to 500 (maximum score : severe).
To evaluate the proportion of responders according to the European Medicines Agency (EMA) definition, after 8 weeks of treatment | Day 56 and day 84
  Proportion of responders at D56 and D84 according to the EMA definition (patients with a subject's global assessment of efficacy scale (Irritable Bowel Syndrome - Global Improvement Scale, IBS-GIS) of the highest two improvement grades of a 7-point scale (1 : significantly relieved to 7 : significantly worse), and with an abdominal pain score which has improved at least 30% compared to baseline). The abdominal pain score will be taken from the abdominal pain 11-point NRS.(0 : no pain to 10 : worse possible pain)
Assessment of the safety and tolerability of Saccharomyces boulardii CNCM I-745. Irritable Bowel Syndrome (IBS) patients in comparison to placebo. Recording adverse events | From baseline to day 84
  Safety endpoint : Recording of adverse events and serious adverse events (number of events and number of participants with at least one event)
Assessment of the safety and tolerability of Saccharomyces boulardii CNCM I-745. Irritable Bowel Syndrome (IBS) patients in comparison to placebo. Recording changes in pulse rate | From baseline to day 84
  Safety endpoint : changes in pulse rate (beats per minute)
Assessment of the safety and tolerability of Saccharomyces boulardii CNCM I-745. Irritable Bowel Syndrome (IBS) patients in comparison to placebo. Recording changes in blood pressure | From baseline to day 84
  Safety endpoint : changes in blood pressure (millimeter of mercury (mmHg))
Assessment of the safety and tolerability of Saccharomyces boulardii CNCM I-745. Irritable Bowel Syndrome (IBS) patients in comparison to placebo. Recording changes in body weight | From baseline to day 84
  Safety endpoint : changes in body weight (kilograms (kg))

OTHER OUTCOMES:
To explore the proportion of responders in Irritable Bowel Syndrome - with predominant Diarrhea (IBS-D) subgroup, according to the US Food and Drug Administration (FDA) definition. | Day 56 and day 84 compared with baseline
  Proportion of responders in Irritable Bowel Syndrome - with predominant Diarrhea (IBS-D) subgroup (Rome IV criteria at inclusion), according to the FDA definition (≥30% improvement in abdominal pain and a ≥50% reduction in number of days per week with at least one stool that has a consistency of type 6 or 7 on the Bristol Stool Form Scale (BSFS)) at D56 and D84 compared with baseline. The abdominal pain score will be taken from the abdominal pain 11-point numerical rating scale (NRS).
To explore the proportion of patients who improved ≥ 75 points on Irritable Bowel Syndrome Symptom Severity Scale(IBS-SSS). | Day 56 compared to baseline
  Irritable Bowel Syndrome Symptom Severity Scale (IBS-SSS) is a scale evaluating the severity of the disease from 0 (minimum score : not severe) to 500 (maximum score : severe).
To explore the effect of Saccharomyces boulardii CNCM I-745 on each Irritable Bowel Syndrome- Quality of Life (IBS-QOL) subscore in comparison to placebo. | Day 56 and day 84 compared to baseline
  Change from baseline in Irritable Bowel Syndrome- Quality of Life (IBS-QOL)subscores (Dysphoria, Interference with activity, Body Image, Health worry, Food avoidance, Social Reaction, Sexual, and Relationships) at D56 and D84. Minimum score is 0 : poor quality of life. Maximum score : 100 : better quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Oana Bernard, DR, Study Director — Biocodex
Locations (10):
- Portugal (2):
  - Hospital de Braga, Braga
  - Hospital da Luz, Lisbon
- Spain (8):
  - Hospital Universitario Vall d'Hebron, Barcelona
  - Hospital Universitario de León, León
  - Hospital Universitario Gregorio Marañon & Centro de Salud Pavones, Madrid
  - Hospital Clínico San Carlos, Madrid
  - Hospital Universitario La Paz & Hospital Carlos III, Madrid
  - Hospital Universitario Costa del Sol, Marbella
  - Hospital Universitario Regional de Málaga, Málaga
  - Hospital Universitario Central de Asturias & Centro de Salud la Lila, Oviedo